CLINICAL TRIAL: NCT04166734
Title: Pembrolizumab and Hypofractionated Stereotactic Radiotherapy in Patients With Malignant Pleural Mesothelioma
Acronym: MESO-PRIME
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to slow recruitment and insufficient further funding.
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CCR4583
Record Dates: First submitted 2019-11-08; First posted 2019-11-18 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Advanced Malignant Pleural Mesothelioma
Keywords: Advanced malignant pleural mesothelioma; mesothelioma; pembrolizumab; radiotherapy; SBRT; External Beam Stereotactic Body Radiotherapy
MeSH Terms: conditions — Mesothelioma | interventions — pembrolizumab; Radiosurgery

STUDY DESIGN:
Intervention Model Description: Initial safety phase followed by an Expansion phase
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Initial safety cohort (Other): Patients will receive an initial dose of pembrolizumab in week 1 dosed at 200 mg. They will then receive SBRT dosed at 30 Gy in 3 fractions (#) alternate days in week 3. Treatment with pembrolizumab will be continued dosed at 200 mg given every 3 weeks.
  Interventions: Drug: Pembrolizumab; Radiation: Stereotactic Body Radiotherapy (SBRT)
- Expansion cohort (Other): An additional 12 patients will be recruited for this cohort. Patients will receive an initial dose of pembrolizumab at 200 mg in week 1. This will be followed in by SBRT dosed at 30 Gy in 3 fractions (#) alternate days in week 3. Treatment with pembrolizumab will be continued dosed at 200 mg given every 3 weeks.
  Interventions: Drug: Pembrolizumab; Radiation: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab will be continued dosed at 200 mg given every 3 weeks
  Drug: Pembrolizumab Pembrolizumab in week 1 dosed at 200 mg (prior to SBRT) and then treatment with pembrolizumab will be continued dosed at 200 mg given every 3 weeks.
  Other Names: Keytruda
Radiation: Stereotactic Body Radiotherapy (SBRT) — Stereotactic Body Radiotherapy (SBRT) 30 Gy 3 fractions (#)
  Other Names: SBRT

SUMMARY:
This is a multi-centre non-randomised open-label phase 1 trial of pembrolizumab given in combination with SBRT to part of a pleural-based lesion in patients with unresectable MPM. This study will recruit up to 18 patients whose MPM has progressed beyond first-line of palliative chemotherapy, with a platinum-based doublet, and now requires further palliative systemic treatment, or have declined first-line palliative chemotherapy, however must have been considered suitable for a platinum doublet chemotherapy.

DETAILED DESCRIPTION:
The study will be conducted in two parts; an initial safety phase (Part A), followed by an expansion cohort (Part B). The initial safety phase (Part A) is based on a 3+3 design such that patients will be treated in a cohort of 3-6 patients. A maximum of 6 patients will be allocated to Part A exploring SBRT 30 Gy in 3 fractions in combination with pembrolizumab. If there is more than one DLT in the first 3 patients or two or more DLTs in the first 6 patients, this treatment combination will be deemed as being unacceptable and it would lead to termination of the study. During the expansion cohort (Part B), 12 patients will have SBRT 30 Gy in 3 fractions with pembrolizumab to obtain additional safety and response data. Maintenance pembrolizumab will continue until disease progression, unacceptable toxicities, the patient withdraws consent to the trial, or the patient has completed 35 cycles of treatment. A maximum of 18 patients will be treated in the study.

All patients will receive pembrolizumab on cycle (C) 1 day (D) 1, in Part A and B of the study. All patients will receive SBRT on C1D15, C1D17 and C1D19, as per SBRT protocol. Patients in part A will receive SBRT 30 Gy in 3#. Patients in Part B will receive 30 Gy in 3 fractions if considered safe after part A. All patients in Part A and Part B will receive pembrolizumab dosed at 200 mg every 3 weeks, until disease progression, unacceptable toxicities, the patient withdraws consent from the trial or the patient has completed 35 cycles of treatment.

In the initial safety cohort, a minimum of 3 patients will be treated at the SBRT dose of 30Gy in 3 fractions combined with pembrolizumab. The gap left between the treatments of each subsequent patient will start after the second cycle of Pembrolizumab in the previous dosed patient to mitigate against multiple patients suffering from acute toxicity. The DLT period for this study is 12 weeks from the last dose of SBRT (i.e. at C6D1). Patients included in Part A will be considered by the Safety Review Committee (SRC) once the 3rd and 6th patient in the Part A cohort has completed the DLT period. If 0 out of 3 patients experience a DLT, or if 1 out of 3 patients experience a DLT in Part A, then the cohort will be expanded to 6 patients. If 1 in 6 patients experience a DLT, then it will be acceptable to move forward to the expansion cohort (Part B).

However, if ≥ 2 in 6 patients (or more than 1 in the first 3 patients) experience a DLT then the maximum administered dose (MAD) will have been reached. If the MAD is seen at a dose level of 30 Gy in 3# then the study will be terminated.

While waiting for 3 or 6 patients to complete the DLT period, no additional patients will be recruited. Further patients can only be recruited after the SRC has reviewed the toxicity data for the cohort to proceed to Part B. Patients obtaining complete response or having completed 35 cycles of pembrolizumab must discontinue and may recommence for additional 17 cycles upon subsequent disease, the CI/PI will need to discuss with the sponsor and MSD, on a case by case basis for the continuation of pembrolizumab

ELIGIBILITY:
Inclusion Criteria:

1. Patients should be ≥18 years old on the day of signing the informed consent.
2. Patients must have a histological or cytological diagnosis of MPM.
3. Patients should have non-radically treatable MPM (i.e. not being considered for extrapleural pneumonectomy or pleurectomy and decortication).
4. Patients must have measurable disease as assessed by mRECIST (i.e. at least a 1 cm rind of MPM at 2 sites on 3 different levels).
5. Patients must have had disease progression or be intolerant of standard first-line palliative chemotherapy for MPM. Patients who have declined first-line palliative chemotherapy must have been suitable for platinum-doublet combination chemotherapy.
6. Patient should have an ECOG performance status 0-1.
7. Patients should be able to tolerate a course of stereotactic radiotherapy as assessed by the investigator.
8. Patients should have pleural based disease, away from critical structures, and suitable for treatment to part of lesion with SBRT for pleural mesothelioma.
9. Patients must have adequate organ function including MRC dyspnoea score <3 and adequate baseline lung function tests, with an FEV1 > 0.8L or >30% of predicted and a TLCO > 30%.
10. Demonstrate adequate organ function (based on bloods within 10 days of C1D1).
11. Have provided tissue from an archival tissue sample or newly obtained tissue sample.
12. Female patient of childbearing potential should have a negative serum pregnancy within 72 hours prior to receiving the first dose of study medication (C1D1). Female patients of childbearing potential should be willing to use highly effective methods of contraception for the course of the study through 120 days after the last dose of study medication. Female of childbearing potential is defined as women following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
13. Male patients should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
14. Be willing to provide informed consent for the trial.

Exclusion criteria

1. Patients who have taken any investigational medicinal product or have used an investigational device within 4 weeks of the first dose of pembrolizumab. Patients are allowed to participate in additional observational studies.
2. Patients who have received prior chemotherapy, targeted small molecule therapy or radiotherapy within 4 weeks prior to the first dose of pembrolizumab.
3. Patients with a diagnosis of immunodeficiency or be receiving systemic steroid therapy (>7.5 mg of prednisone / >1 mg of dexamethasone or their equivalent dose) or any other form of immunosuppressive therapy within 7 days prior to the first dose.
4. Patients with evidence of active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents or an autoimmune disease that is currently quiescent off any treatment, but deemed at risk of a significant flare if treated on this protocol.
5. Patients who have received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
6. Patients with evidence of active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided the brain metastases are stable and there is no evidence of new or enlarging brain metastases.
7. Patients who have had previous radiotherapy to the thorax or other neighbouring region that would preclude the safe administration of SBRT for MPM.
8. Patients with evidence of interstitial lung disease or active, non-infectious pneumonitis.
9. Patients with evidence of additional malignancy that is progressing or requires active treatment.
10. Patients with a history or current evidence of any condition, therapy, or laboratory abnormality that might confound trial results, interfere with the patient's participation or is not in the best interest of the patient.
11. Patients with psychiatric or substance abuse disorders that would interfere with patients participation.
12. Patients who are pregnant / breastfeeding or expecting to conceive within the duration of the trial, starting with the screening visit through 120 days after the last dose.
13. Patients with a history of HIV, HIV 1/2 antibodies, Hepatitis B or Hepatitis C.
14. Patients with any active infection requiring systemic treatment
15. Patients who have received a live vaccine within 30 days prior to the first dose of trial treatment.
16. Patients with known hypersensitivity to the active substance pembrolizumab or to any of the excipients listed in the IB.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fiona McDonald, Study Chair — Royal Marsden NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Royal Marsden NHS Foundation Trust, Chelsea
  - Beatson West of Scotland Cancer Centre, Glasgow

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of five participants were recruited to the trial, all to the initial safety cohort. The participants were registered between February 2021 and March 2022.
Groups:
- Initial Safety Cohort: Patients will receive an initial dose of pembrolizumab in week 1 dosed at 200 mg. They will then receive SBRT dosed at 30 Gy in 3 fractions (#) alternate days in week 3. Treatment with pembrolizumab will be continued dosed at 200 mg given every 3 weeks.
  Pembrolizumab: Pembrolizumab will be continued dosed at 200 mg given every 3 weeks
  Drug: Pembrolizumab Pembrolizumab in week 1 dosed at 200 mg (prior to SBRT) and then treatment with pembrolizumab will be continued dosed at 200 mg given every 3 weeks.
  Stereotactic Body Radiotherapy (SBRT): Stereotactic Body Radiotherapy (SBRT) 30 Gy 3 fractions (#)
- Expansion Cohort: An additional 12 patients will be recruited for this cohort. Patients will receive an initial dose of pembrolizumab at 200 mg in week 1. This will be followed in by SBRT dosed at 30 Gy in 3 fractions (#) alternate days in week 3. Treatment with pembrolizumab will be continued dosed at 200 mg given every 3 weeks.
  Pembrolizumab: Pembrolizumab will be continued dosed at 200 mg given every 3 weeks
  Drug: Pembrolizumab Pembrolizumab in week 1 dosed at 200 mg (prior to SBRT) and then treatment with pembrolizumab will be continued dosed at 200 mg given every 3 weeks.
  Stereotactic Body Radiotherapy (SBRT): Stereotactic Body Radiotherapy (SBRT) 30 Gy 3 fractions (#)
Period: Overall Study
Arm/Group | Initial Safety Cohort | Expansion Cohort
Started | 5 | 0
Commenced Pembrolizumab | 5 | 0
Completed 30Gy SBRT in 3 Fractions | 5 | 0
Completed 35 Cycles Pembrolizumab | 0 | 0
Completed | 0 | 0
Not Completed | 5 | 0
Not completed — Lack of Efficacy | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Intercurrent illness | 1 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: All patients treated with at least one dose of trial treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Initial Safety Cohort | Expansion Cohort | Total
Number analyzed (Participants) | 5 | 0 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 2 |  | 2
  >=65 years | 3 |  | 3
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 72 [62 to 76] |  | 72 [62 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 3 |  | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian (white) | 5 |  | 5
Region of Enrollment [Number; unit: participants]
  United Kingdom | 5 |  | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Dose Limiting Toxicity (DLT)
Description: Dose limiting toxicity is assessed using CTCAE v5.0 and defined as any one of: neutropenia with fever grade>=3; neutropenia grade>=4; thrombocytopenia with bleeding grade >=3; thrombocytopenia grade >=4; any non-haematological toxicity grade >=3 which is definitely, probably or possibly related to the combination of pembrolizumab and SBRT
Time Frame: Worst grade as assessed at cycle 1 day 1 of pembrolizumab, at each of three radiotherapy fractions (cycle 1 days 15, 17, 19) and then at day 1 of each 21 day cycle, up to 12 weeks from last dose of SBRT (i.e. cycle 6 day 1)
Population: Patients who remained on trial for the duration of the DLT time frame
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Safety Cohort | Expansion Cohort
Number analyzed (Participants) | 3 | 0
Participants | 0 |

2. Secondary Outcome: Worst Acute Toxicity Grade
Description: Number of patients by worst recorded grade of acute toxicity, assessed using CTCAE v5.0
Time Frame: as for outcome 1
Population: All patients who received at least one dose of trial treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Safety Cohort | Expansion Cohort
Number analyzed (Participants) | 5 | 0
Participants
  Max grade 3 | 3 | 0
  Max grade 2 | 2 |

3. Secondary Outcome: Overall Response Rate
Description: Proportion of patients with best recorded response as assessed using RECIST v1.1 of complete or partial response
Time Frame: Response assessed from start of pembrolizumab, every 9 weeks for the first 6 months, then every 12 weeks thereafter, until the first instance of documented disease progression, start of new anti-cancer treatment, death or end of study (24 months)
Population: All patients who commenced trial treatment and who were assessed at least once for response
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Safety Cohort | Expansion Cohort
Number analyzed (Participants) | 5 | 0
Participants | 1 | 0

4. Secondary Outcome: Disease Control Rate
Description: Proportion of patients with best recorded response as assessed using RECIST v1.1 of complete or partial response or stable disease
Time Frame: as for outcome 3
Population: All patients who commenced trial treatment and who were assessed at least once for response
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Safety Cohort | Expansion Cohort
Number analyzed (Participants) | 5 | 0
Participants | 3 | 0

5. Secondary Outcome: Overall Survival (OS) at Six Months
Description: Proportion of patients alive at six months
Time Frame: 6 months after start of pembrolizumab treatment
Population: All patients who commenced trial treatment and did not withdraw before 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Safety Cohort | Expansion Cohort
Number analyzed (Participants) | 3 | 0
Participants | 3 | 0

6. Secondary Outcome: Overall Survival (OS) at Twelve Months
Description: Proportion of patients alive at twelve months
Time Frame: 12 months after start of pembrolizumab treatment
Population: All patients who commenced trial treatment and did not withdraw before 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Safety Cohort | Expansion Cohort
Number analyzed (Participants) | 3 | 0
Participants | 2 |

7. Secondary Outcome: Progression Free Survival at 6 Months
Description: Proportion of patients alive and free from progression at six months
Time Frame: 6 months after commencing pembrolizumab treatment
Population: Patients who commenced trial treatment and did not withdraw before progression and before 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Safety Cohort | Expansion Cohort
Number analyzed (Participants) | 4 | 0
Participants | 2 | 0

8. Secondary Outcome: Progression Free Survival at 12 Months
Description: Proportion of patients alive and free from progression at twelve months
Time Frame: 12 months after commencing pembrolizumab treatment
Population: Patients who commenced trial treatment and did not withdraw before progression and before 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Safety Cohort | Expansion Cohort
Number analyzed (Participants) | 4 | 0
Participants | 2 |

ADVERSE EVENTS:
Time Frame: AEs will be graded and recorded from confirmation of entry into the trial, at cycle 1 day 1 of pembrolizumab, at each of three radiotherapy fractions (cycle 1 days 15, 17, 19) and then at day 1 of each 21 day cycle, until the patients final safety follow up at 30 days after their last dose of pembrolizumab (up to 10 months). All cause mortality is recorded until death or end of trial (24 months).
Description: Adverse events were assessed using CTCAE v5.0. Disease progression of the cancer under study is not considered an AE unless the investigator considers it to be IMP-related or it results in hospitalisation or prolongs existing in-patient hospitalisation or death.
Arm/Group | Initial Safety Cohort | Expansion Cohort
All-Cause Mortality (participants affected / at risk) | 2/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 3/5 | 0/0
Other Adverse Events (participants affected / at risk) | 5/5 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Safety Cohort (N=5) | Expansion Cohort (N=0)
Constipation (Gastrointestinal disorders) | 1 (1) | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | NA
Alanine aminotransferase increased (Investigations) | 1 (1) | NA
Aspartate aminotransferase increased (Investigations) | 1 (1) | NA
Lung infection (Infections and infestations) | 1 (1) | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Safety Cohort (N=5) | Expansion Cohort (N=0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | NA
Lethargy (Nervous system disorders) | 3 (4) | NA
Weight loss (Investigations) | 3 (4) | NA
Alanine aminotransferase increased (Investigations) | 2 (4) | NA
Anorexia (Metabolism and nutrition disorders) | 2 (2) | NA
Aspartate aminotransferase increased (Investigations) | 2 (4) | NA
Constipation (Gastrointestinal disorders) | 2 (2) | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4) | NA
Diarrhea (Gastrointestinal disorders) | 2 (2) | NA
Fatigue (General disorders) | 2 (3) | NA
Fever (General disorders) | 2 (2) | NA
Alkaline phosphatase increased (Investigations) | 1 (1) | NA
Anemia (Blood and lymphatic system disorders) | 1 (1) | NA
Anxiety (Psychiatric disorders) | 1 (1) | NA
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (3) | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | NA
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | NA
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2) | NA
Dry mouth (Gastrointestinal disorders) | 1 (1) | NA
Dysphagia (Gastrointestinal disorders) | 1 (1) | NA
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1) | NA
Flu like symptoms (General disorders) | 1 (1) | NA
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | NA
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | NA
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1) | NA
Hypertension (Vascular disorders) | 1 (4) | NA
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | NA
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | NA
Investigations - other, increased C-reactive protein (Investigations) | 1 (1) | NA
Investigations - other, increased lactate (Investigations) | 1 (1) | NA
Insomnia (Psychiatric disorders) | 1 (1) | NA
Lung infection (Infections and infestations) | 1 (1) | NA
Lymphocyte count decreased (Investigations) | 1 (1) | NA
Papilledema (Eye disorders) | 1 (1) | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | NA
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 (1) | NA
Vomiting (Gastrointestinal disorders) | 1 (1) | NA
Investigations - other, raised urea (Investigations) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT04166734/Prot_000.pdf